CLINICAL TRIAL: NCT06028373
Title: A First-in-Human Phase I Study of ATG-031 in Patients With Advanced Solid Tumors or B-cell Non-Hodgkin Lymphomas
Brief Title: A Study of ATG-031 in Advanced Solid Tumors or B-cell Non-Hodgkin Lymphomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Antengene Biologics Limited (Industry)
Responsible Party: Sponsor
Organization: Antengene Corporation (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ATG-031-001
Record Dates: First submitted 2023-08-25; First posted 2023-09-08 (Actual); Last update posted 2025-06-09 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumors; B-cell Non-Hodgkin Lymphomas
Keywords: ATG-031; solid tumor; CD 24

STUDY DESIGN:
Intervention Model Description: Dose levels are 0.03 mg/kg、 0.1 mg/kg、0.3 mg/kg 、0.5mg/kg ,or other dose level less than 1.0mg/kg determined by SRC
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- ATG-031 dose level 1 (Active Comparator): Patients with advanced solid tumors or B-cell non-Hodgkin lymphomas will be enrolled in the Dose-Escalation Phase.
  Dose level is 0.03 mg/kg
  Interventions: Drug: ATG-031
- ATG-031 dose level 2 (Active Comparator): Patients with advanced solid tumors or B-cell non-Hodgkin lymphomas will be enrolled in the Dose-Escalation Phase.
  Dose level is 0.1 mg/kg
  Interventions: Drug: ATG-031
- ATG-031 dose level 3 (Active Comparator): Patients with advanced solid tumors or B-cell non-Hodgkin lymphomas will be enrolled in the Dose-Escalation Phase.
  Dose level is 0.3 mg/kg
  Interventions: Drug: ATG-031
- ATG-031 dose level 4 (Active Comparator): Patients with advanced solid tumors or B-cell non-Hodgkin lymphomas will be enrolled in the Dose-Escalation Phase.
  Dose level is 1.0 mg/kg
  Interventions: Drug: ATG-031
- ATG-031 dose level 5 (Active Comparator): Patients with advanced solid tumors or B-cell non-Hodgkin lymphomas will be enrolled in the Dose-Escalation Phase.
  Dose level is 2.0 mg/kg
  Interventions: Drug: ATG-031
- ATG-031 dose level 6 (Active Comparator): Patients with advanced solid tumors or B-cell non-Hodgkin lymphomas will be enrolled in the Dose-Escalation Phase.
  Dose level is 4.0 mg/kg
  Interventions: Drug: ATG-031
- ATG-031 dose level 7 (Active Comparator): Patients with advanced solid tumors or B-cell non-Hodgkin lymphomas will be enrolled in the Dose-Escalation Phase.
  Dose level is 6.0 mg/kg
  Interventions: Drug: ATG-031
- ATG-031 dose level 8 (Active Comparator): Patients with advanced solid tumors or B-cell non-Hodgkin lymphomas will be enrolled in the Dose-Escalation Phase.
  Dose level is 9.0 mg/kg
  Interventions: Drug: ATG-031

INTERVENTIONS:
Drug: ATG-031 — ATG-031 will be infused Q3W on Day 1 of each cycle, at the starting dose of 0.03 mg/kg and a maximum dose of 9 mg/kg in the Dose Escalation Phase, and the defined MTD if available or OBD in the Dose Expansion Phase. Based on the emerging PK, PDx, safety, and other relevant data, SRC may decide to explore alternative dosing schedules.

SUMMARY:
ATG-031 study (alias: PERFORM) is a multicenter, open-label, Phase 1 study of ATG-031 in patients with advanced solid tumors or B-NHL. The study design includes a Dose Escalation Phase and a Dose Expansion Phase, and will enroll patients with advanced solid tumors (i.e., preferred tumor types) or relapsed/refractory (R/R) B-NHLs. The study's primary objective is to evaluate the safety and tolerability of ATG-031 and determine the RP2D（Refered Phase II dose） of ATG-031.

DETAILED DESCRIPTION:
This is a multicenter, open-label, Phase 1 study of ATG-031 in patients with advanced solid tumors or B-NHL. The study design includes a Dose Escalation Phase and a Dose Expansion Phase. Dose Escalation Phase: approximately 30-48 patients . Dose Expansion Phase: the number of patients enrolled will depend on the number of disease cohorts to be expanded and data observed in the Dose Escalation Phase.The Dose Escalation Phase will enroll patients with advanced solid tumors. Based on data from dose escalation (e.g., adverse events [AEs], dose-limiting toxicity [DLT], efficacy data, pharmacodynamic [PDx] data, or pharmacokinetic [PK] data), the Dose Expansion Phase will enroll patients with selected advanced solid tumors or B-NHL.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histological or cytologically confirmed advanced solid tumor or B-NHL which have relapsed from or been refractory to all locally available standard therapies.
2. Adequate hepatic function:

   1. AST and ALT ≤ 2.5×times ULN (≤ 5 × ULN if liver metastases).
   2. Total bilirubin ≤ 1.5×ULN (except Gilbert syndrome).
   3. Lipase and amylase ≤ 2×ULN.
3. Adequate renal function: calculated creatinine clearance of ≥ 40 mL/min using the Cockroft- Gault formula.
4. Adequate bone marrow function without growth factors or blood transfusion within 7 days of the first dose of study treatment.

   1. Absolute neutrophil count (ANC) ≥ 1.5×109/L.
   2. Platelet count ≥ 100×109/L.
   3. Hemoglobin ≥ 90 g/L.

Key Exclusion Criteria:

1. Patients with CNS malignancies, except those who are clinically stable for ≥ 4 weeks and off corticosteroids following prior surgery, whole-brain radiation, or stereotactic radiosurgery.
2. Received any other investigational product or prior systemic anticancer therapy including chemotherapy, immunotherapy, radiotherapy, or other anticancer within 21 days prior to first dose of study
3. Grade ≥3 irAEs or irAEs that lead to discontinuation of prior immunotherapy.8. Other primary malignancies developed within 5 years prior to the first dose of the study treatment
4. Other primary malignancies developed within 5 years prior to the first dose of the study treatment
5. Have active or previous autoimmune diseases that are likely to recur or are at risk of such diseases judged by the investigator.
6. Major cardiovascular disease
7. Active hepatitis B and/or hepatitis C (HBV-DNA or HCV-RNA detectable by local laboratory, respectively).
8. Patients with history of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
9. A history of allograft organ transplantation for solid tumor or allogeneic hematopoietic stem cell transplantation for B-NHL patients).
10. Patients who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
AE | 90 days after last dose of treatment
  Evaluate the safety and tolerability of ATG-031
DLT | at the end of cycle 2 ( each cycle is 21 days)
  Evaluate the safety and tolerability of ATG-031
RP2D | at the end of dose escalation, about 1 year
  RP2D will be determined based on safety, tolerability, PK, and preliminary efficacy data

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of California San Francisco (UCSF), San Francisco, California
  - Regents of the University of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas